CLINICAL TRIAL: NCT01750580
Title: A Phase 1 Study of BMS-986015, an Anti-KIR Monoclonal Antibody, Administered With Ipilimumab, an Anti-CTLA4 Monoclonal Antibody, in Subjects With Select Advanced Solid Tumors
Brief Title: Safety Study of BMS-986015 (Anti-KIR) in Combination With Ipilimumab in Subjects With Selected Advanced Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA223-002
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: CANCER, NOS
MeSH Terms: conditions — Neoplasms | interventions — lirilumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: Lirilumab + Ipilimumab (Experimental): Lirilumab and Ipilimumab on specific days
  Interventions: Drug: Lirilumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Lirilumab
  Other Names: BMS-986015; IPH-2102; ANTI-KIR
Drug: Ipilimumab
  Other Names: BMS-734016

SUMMARY:
To assess the safety and tolerability, characterize the dose-limiting toxicities (DLTs), and identify the maximally tolerated dose (MTD) of BMS-986015 given in combination with ipilimumab in subjects with select advanced (metastatic and/or unresectable) solid tumors.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Histologic confirmation of one of the following solid tumors that is advanced (unresectable or metastatic) for dose escalation or cohort expansion:Non-Small Cell Lung Cancer (NSCLC), Castrate Resistant Prostate Cancer (CRPC), Melanoma (MEL)
* At least one measurable lesion at baseline by Computed tomography (CT) or Magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Biopsies: Subjects in the melanoma cohort must have at least 1 tumor site that can be biopsied at acceptable clinical risk
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Estimated life expectancy of ≥ 12 weeks
* White blood cell (WBC) ≥2000/μL, Neutrophils ≥1500/μL, Platelets ≥ 100x1000/μL, Hemoglobin ≥ 8.5 g/dL, creatinine ≤ 1.5 X upper limit of normal (ULN) mL/min, Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 3x ULN
* Normal thyroid function or be on stable hormone supplementation

Exclusion Criteria:

* Participation in any prior clinical study with BMS-936558 or ipilimumab that has overall survival listed as a primary/co-primary endpoint
* Subjects with known or suspected brain metastasis
* Subjects with active autoimmune disease, uncontrolled or significant cardiovascular disease
* Prior therapy with anti- Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) antibody or anti- Killer cell immunoglobulin-like receptor (KIR) antibody
* Grade 2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the rate of adverse events, and serious adverse events | Approximately 510 days

SECONDARY OUTCOMES:
Efficacy as measured by tumor assessment | Assessed from the start of treatment (ay 1) to the end of treatment (week 60) and for 90 days in follow-up
The maximum observed serum concentration (Cmax) of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2. (EOI is end of infusion, EOT is end of treatment
The time of maximum observed serum concentration (Tmax) of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2
Area under the serum concentration-time curve in one dosing interval [AUC(TAU)] of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, EOT, follow-up 1 and follow-up 2
Apparent total body clearance (CL) of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2
Apparent volume of distribution at steady state (Vss) of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2
Serum half-life (T-HALF) of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2
Trough observed serum concentration (Cmin) of BMS-986015 and Ipilimumab | up to 18 timepoints following each dose during Weeks 1, (0h, EOI and 24h), 2, 3, 4, 10, (0h, EOI and 24h), 11, 13, 24, (0h and EOI), 36, 48, 60, follow-up 1 and follow-up 2
Immunogenicity as measured by the incidence of Ipilimumab and anti-Killer cell immunoglobulin-like receptor (KIR) (BMS-986015) anti-drug antibodies (ADA) | up to 11 timepoints during Weeks 1, 3, 4, 10, 13, 24, 36,48, 60, follow-up 1 and follow-up 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University Of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx